CLINICAL TRIAL: NCT02798965
Title: Prevalence of Circulating Parvovirus Genome in Recently Diagnosed Graves' Disease: a Case-control Study
Acronym: GPCBasedow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AOL10-DR-DESAILLOUD
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Graves Disease
Keywords: parvovirus genome
MeSH Terms: conditions — Graves Disease | interventions — Serologic Tests

ARMS (2):
- Control (Other): patients with goiter or nodule
  Interventions: Biological: serodiagnosis
- Graves' disease (Experimental): patients with Graves' disease
  Interventions: Biological: serodiagnosis

INTERVENTIONS:
Biological: serodiagnosis

SUMMARY:
Lymphocytic thyroiditis is the most common autoimmune disease, usually affecting young women. Although the aetiology and pathogenesis remain obscure, the most widely accepted hypothesis is an interaction between a genetic predisposition and an environmental trigger factor such as viral infection. Parvovirus infections have been proposed as trigger factors for Hashimoto's thyroiditis and Graves' disease.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease :patients treated for Graves' disease, the diagnosis date less than 4 months
* Control : patients cared for nodules or goiter

Exclusion Criteria:

* Patients undergoing immunosuppressive therapy including corticosteroids

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
prevalence of circulating parvovirus genome | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Rachel DESAILLOUD, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] https://www.em-consulte.com/article/753902/detection-de-levb19-parvovirus-b19-dans-les-thyroc